CLINICAL TRIAL: NCT03597737
Title: Utility of an APP for the Monitoring of Irruptive Oncological Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OncoApp
Record Dates: First submitted 2018-06-19; First posted 2018-07-24 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Oncology; Pain, Acute; Pain, Chronic
MeSH Terms: conditions — Neoplasms; Acute Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: One condition
Masking Description: Patients will be informed of the condition they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment as usual + APP (Experimental): Participants at this condition will receive the usual medical treatment for their pain but also they will be monitored daily using the Pain Monitor APP. Alarms will be generated in the face of certain preestablished events. Physicians will be asked to call patients and change/stop treatment if an alarm is received.
  Interventions: Device: Pain APP

INTERVENTIONS:
Device: Pain APP — pain app Pain Monitor app has been developed by a multidisciplinary pain expert panel, including physicians, psychologists, and nurses. Content has been validated in a previous study and usability has been shown to be excellent.

SUMMARY:
The present investigation aims at exploring the effect of including a pain app called Pain Monitor irruptive oncological pain for chronic pain patients' daily monitoring. Two conditions will be set:

1. usual treatment (waiting list)
2. usual treatment + APP

DETAILED DESCRIPTION:
Irruptive oncological pain (IOP) is defined as an exacerbation of pain in cancer patients whose base pain is stable (e.g., less than 4 on a scale of 0 to 10 for more than 12 hours a day) and is well controlled with opioids. This pain increase can appear both spontaneously and associated to a specific determining factor, be it predictable or unpredictable. The IOP tends to appear quickly (3-5 minutes) and usually have a short duration (average 30 minutes, although pain may last more than 60 minutes) and moderate intensity to elevated . The median episodes of breakthrough pain per day is of 3.

The prevalence of IOP is alarmingly high. A review study of 19 works scientists places the number of cancer patients with IOP in approximately 60%. In addition, the IOP is associated with a significant decrease in the quality of life of the patients. For example, a study conducted in different countries in Europe with 1000 cancer patients revealed that in more than 80% of the participants, the appearance of breakthrough pain completely interrupted their activities. Only 11% of the patients interviewed expressed that the IOP did not interfere in their activities. For the rest of the patients, the most affected areas were sleep and emotional well-being. In addition to these costs in the quality of life of patients with IOP, recent studies have warned of the consequences of this type of pain. Thus, an investigation carried out in the United States evidenced that three quarters of the patients interviewed had experienced important economic losses as a result of the pain, being the average direct costs associated with the IOP of $ 891 per person per month.

Aiming to choose the most appropriate study methodology for this type of pain (often unpredictable and of short duration), the investigators have reviewed the works carried out up to the moment on characteristics and treatment of the IOP. Descriptive studies on IOP tend to use a most retrospective observational methodology, which can lead to biases and inaccuracies. For example, in the most ambitious study carried out so far, 1000 patients with IOP were urged to remember the characteristics of pain episodes, such as the average intensity, the approximate average duration and the average number of events per day.

Regarding the investigations on the effectiveness of the treatment of the IOP, the studies comparing different drugs tend to perform clinical trials, while to study the response to a particular drug, seems more adequate continuous assessment of each patient during an IOP episode. This last methodology with repeated measures seems the most adequate in IOP, since the use of clinical trials with few measures (baseline, post-treatment and follow-up) has the limitation of not allowing daily monitoring of patient's pain episodes.

Although daily assessments seems to be the most suitable design for the monitoring of patients with IOP, the implementation of this type of methodology could be very expensive because requires continuous evaluation. To facilitate this, several studies have already shown that mobile applications (APP) can effectively monitor the evolution of a wide range of pathologies in the context of health. In fact, a controlled clinical study recently made found that the records eco-friendly through mobile APPs were more reliable than registers with pencil and paper.

As for the existing APPs in pain, an exhaustive review of the available APPs revealed that there was little evidence to support the use of these technologies. Specifically, these authors showed that the most APPs did not specify whether their content was validated, APPs did not include psychological components and none had been applied in a clinical study. In the light of these results, the investigators contacted the Labpsitec research team of the University Jaume I, who have developed and validated a pain application called "Pain Monitor".

The APP daily evaluates the variables recommended by the Initiative on Methods, Measurement and Evaluation of Pain (IMMPACT): intensity of the pain, use of rescue analgesics, pain interference in functioning, state of mood, general perception of health and evaluation of treatment effectiveness. In addition, "Pain Monitor" also assesses psychological factors and behavior that influence the experience of pain: catastrophism, acceptance, fear / avoidance and coping. The APP seems especially indicated for IOP monitoring since, following the recommendations of the guide "Comprehensive approach to the patient with irruptive oncological pain", allows patients access at any time to record the characteristics of pain (place, intensity, duration and characteristics of pain) and frequency of use of medication for the spikes of pain. Finally, the APP allows to create alarms so that, undesirable clinical events (e.g., severe or recurrent adverse effect, increased pain basal, no pain reduction after use of rescue medication, low adherence to treatment), are sent by email to the principal investigator of the study.

Thus, the study objective is to test if the introduction of the Pain Monitor APP in the day-to-day work of the pain unit improves pain management of irruptive oncological pain patients. To do this, it is necessary to compare the evolution of patients who follow the usual treatment at the pain unit (without app) with a group of patients who do use the Pain Monitor APP.

The investigators will perform a clinical trial comparing the 2 conditions mentioned above:

1. usual treatment (waiting list)
2. usual treatment + APP

Therefore, this is a clinical trial without drugs. This is not an observational study since the physicians of patients in the app + alarms condition will be asked to react to an alarm (i.e., if the patient has nausea for 3 consecutive days) by calling the patient and changing the treatment telematically, if necessary, so that the patient can collect the prescription at his primary care center. If the condition APP results in a better treatment of irruptive oncological pain patients, participants of the waiting list will be offered the possibility to use the app at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* The patient is over 18 years of age
* Irruptive oncological pain
* The patient has a mobile phone with Android operating system
* The patient has the physical ability to use the application
* The patient does not present psychological and / or cognitive alterations or problems with language that make their participation difficult- The patient voluntarily wants to participate and signs the informed consent

Exclusion Criteria:

* The patient is under 18 years
* The patient does not have a mobile phone or has a mobile phone in which Android is not the operating system (the app is currently only available for Android for economic reasons)
* The patient does not have the physical capacity to use the application
* The patient does not have the capacity to participate due to psychological and / or cognitive alterations or problems with language
* The patient does not want to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
Change in average pain intensity in the past week assessed by a Numerical Rating Scale in the Brief Pain Inventory-Short Form | Twice (first day of study and 30 days after, at the end of study)
  The Brief Pain Inventory-Short Form (BPI-SF) will be used to measure average pain intensity. The item has a response range from 0 (no pain) to 10 (pain as bad as you can imagine). Higher scores represent higher pain intensity levels
Change in side effects of pain medication | Twice (first day of study and 30 days after, at the end of study)
  A list of the most frequent side effects of pain medication has been created. Responses are dichotomous (0=did not experience the side effect; 1=experienced the side effect)

SECONDARY OUTCOMES:
Change in depression measured by the Sadness scale in the POMS | Twice (first day of study and 30 days after, at the end of study)
  The Profile of Mood States (POMS) questionnaire will be used to measure mood. The questionnaire includes 30 items that describe how the participant feels. For this outcome depression scale (5 items) will be used. Each item has a response range from 0 (not at all) to 4 (extremely). Total score ranges from 0 to 20, higher scores represent a worse outcome
Change in anxiety measured by the Tension scale in the POMS | Twice (first day of study and 30 days after, at the end of study)
  The Profile of Mood States (POMS) questionnaire will be used to measure mood. The questionnaire includes 30 items that describe how the participant feels. For this outcome anxiety scale (5 items) will be used. Each item has a response range from 0 (not at all) to 4 (extremely). Total score ranges from 0 to 20, higher scores represent a worse outcome
Change in the amount of rescue medication used in the past week | Twice (first day of study and 30 days after, at the end of study)
  An item exploring the use of rescue medication in the past week has been created. Responses are numerical (the amount of rescue medication is indicated by participants)
Change in average interference of pain in functioning in the past week measured by a Numerical Rating Scale in the Brief Pain Inventory-Short Form | Twice (first day of study and 30 days after, at the end of study)
  The Brief Pain Inventory-Short Form (BPI-SF) will be used to measure pain interference. This questionnaire lists four questions regarding pain intensity and seven regarding pain interference. For this outcome pain interference items will be used. Each item has a response range from 0 (no pain) to 10 (pain as bad as you can imagine). Total score ranges from 0 to 70, higher scores represent a worse outcome
Change in physical health status measured with the Physical Composite Score in the SF12 | Twice (first day of study and 30 days after, at the end of study)
  12-Item Short-Form Health Survey (SF-12) will be used to measure quality of life. This is a questionnaire composed of two scales: physical and mental health. Each scale has a 0-100 range, with higher scores indicating better health-related quality of life
Change in mental health status measured with the Mental Composite Score in the SF12 | Twice (first day of study and 30 days after, at the end of study)
  12-Item Short-Form Health Survey (SF-12) will be used to measure quality of life. This is a questionnaire composed of two scales: physical and mental health. Each scale has a 0-100 range, with higher scores indicating better health-related quality of life
Change in neuropathic symptoms | Twice (first day of study and 30 days after, at the end of study)
  Dolour Neuropathique 4 (DN4) questionnaire will be used to measure neuropathic symptoms. It is a questionnaire composed of 10 items. Each item is scored as 0 (no presence of neuropathic symptom) or 1 (presence of neuropathic symptom). Total score ranges between 0 and 10. It is considered that a patient suffers pain with a neuropathic component when answers affirmatively to 4 or more items of the questionnaire DN4

CONTACTS AND LOCATIONS:
Overall Officials: Azucena García-Palacios, PhD, Study Chair — Universitat Jaume I
Locations (1):
- Consorcio Hospitalario Provincial de Castellón, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No
Only the two principal investigators, Dra. García-Palacios and Dr. Ferrer, will be able to access to individual participant data.

REFERENCES:
- [Background] Suso-Ribera C, Castilla D, Zaragoza I, Ribera-Canudas MV, Botella C, Garcia-Palacios A. Validity, Reliability, Feasibility, and Usefulness of Pain Monitor: A Multidimensional Smartphone App for Daily Monitoring of Adults With Heterogenous Chronic Pain. Clin J Pain. 2018 Oct;34(10):900-908. doi: 10.1097/AJP.0000000000000618. PMID 29659375
- [Background] Garcia-Palacios A, Herrero R, Belmonte MA, Castilla D, Guixeres J, Molinari G, Banos RM. Ecological momentary assessment for chronic pain in fibromyalgia using a smartphone: a randomized crossover study. Eur J Pain. 2014 Jul;18(6):862-72. doi: 10.1002/j.1532-2149.2013.00425.x. Epub 2013 Nov 22. PMID 24921074
- [Background] Olorunto WA, Galandiuk S. Managing the spectrum of surgical pain: acute management of the chronic pain patient. J Am Coll Surg. 2006 Jan;202(1):169-75. doi: 10.1016/j.jamcollsurg.2005.08.007. Epub 2005 Oct 19. No abstract available. PMID 16377510
- [Background] Porta-Sales J, Garzon Rodriguez C, Julia Torras J, Casals Merchan M. [Cancer-related breakthrough pain]. Med Clin (Barc). 2010 Jul 17;135(6):280-5. doi: 10.1016/j.medcli.2010.02.008. Epub 2010 May 6. No abstract available. Spanish. PMID 20451223